CLINICAL TRIAL: NCT05575843
Title: Neurostatus-SMARTCARE in Comparison to Standard Neurostatus- EDSS® - a Swiss Multicenter Randomized Cross-over Study
Brief Title: Neurostatus-SMARTCARE in Comparison to Standard Neurostatus-EDSS®
Acronym: SMARTCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Novartis Pharma AG, Basel, Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2022-01294; ko22DSouza
Record Dates: First submitted 2022-09-07; First posted 2022-10-12 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis (MS)
Keywords: Expanded Disability Status Scale (EDSS); Neurostatus; Neurostatus-eEDSS; Research Center for Clinical Neuroimmunology and Neuroscience Basel (RC2NB)
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Multicentre randomized cross-over study: Randomization 1:1 to group A and group B. Group A undergoes first the Neurostatus-EDSS® and afterwards the Neurostatus-SMARTCARE. Group B starts with the Neurostatus-SMARTCARE and finishes with the Neurostatus-EDSS®. At the next visit the reverse order is applied, by the same neurologist and HCP.
Who Masked: Outcomes Assessor
Masking Description: The HCPs and neurologists performing the examinations are blinded to each others' assessment scores and to the results of previous clinical EDSS examinations. The evaluating experts are blinded to the raters' identity until watching an examination video.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): First neurologist, second nurse
  Interventions: Other: Neurostatus-SMARTCARE; Other: Standard Neurostatus-EDSS
- Group B (Other): First nurse, second neurologist
  Interventions: Other: Neurostatus-SMARTCARE; Other: Standard Neurostatus-EDSS

INTERVENTIONS:
Other: Neurostatus-SMARTCARE — The Neurostatus-EDSS is assessed by HCPs while the examination is video-recorded. HCPs underwent extended training. For details of the examination refer to the second section of the detailed description.
Other: Standard Neurostatus-EDSS — The Neurostatus-EDSS is assessed by neurologists while the examination is video-recorded. Neurologists underwent standard training.

SUMMARY:
The Expanded Disability Status Scale (EDSS) is the gold-standard in assessing disability in Multiple Sclerosis (MS). Its current digital form, the Neurostatus-eEDSS®, often serves as primary endpoint in MS clinical trials.

The pandemic revealed the need for telemedical alternatives to the in-clinic assessment. Therefore, Neurostatus-SMARTCARE was developed: A trained and certified non-neurologist Health Care Professional (HCP) examines the patient while the examination is being video-recorded. The stored video allows a neurologist to re-assess the examination at a later point of time. The future application could be in-home visits through HCPs, in decentralized clinical trials as well as in routine care.

In this study, the concordance rate of Neurostatus examinations between neurologists and HCPs is investigated. With a concordance rate significantly higher than 80%, Neurostatus-SMARTCARE by HCPs can be considered equal to the standard Neurostatus-EDSS by neurologists.

DETAILED DESCRIPTION:
In MS, a specific form of the neurological assessment is the gold-standard to evaluate patients' clinical activity and the evolvement of disability over time: the EDSS. The scale was introduced in 1983 by Kurtzke and has been developed further to the "Neurostatus" by Kappos and co-workers for better reproducibility. In 2011 a digital format of the Neurostatus-EDSS was implemented, the Neurostatus-eEDSS®. It often serves as primary endpoint in MS clinical trials.

Neurostatus-eEDSS® organizes the neurological examination into 8 chapters, which are: visual functional system (FS), brainstem FS, pyramidal FS, cerebellar FS, sensory FS, bowel and bladder FS, cerebral FS and ambulation score. The eight chapters are in turn composed of individual elements (subscores) that investigate neurological functions. Thus, the Neurostatus-eEDSS® results in a total of 121 subcores which are synthetized into 7 FS scores and an ambulation score. The result of the 7 FS scores plus the ambulation score is the EDSS step. The best EDSS step score - 0 (zero) - identifies a normal neurologic examination, and the worst score - 10 (ten) - stands for death due to MS. In-between are intervals of 0.5 steps.

The pandemic revealed the need for telemedical alternatives when as well clinical visits as study visits couldn't be continued routinely. Therefore, the Neurostatus-SMARTCARE was developed: A trained and certified non-neurologist Health Care Professional performs the EDSS examination with the patient while the examination is being video-recorded. The stored video allows a neurologist at a later time-point to review and re-assess the examination and to establish his/ her diagnostic and therapeutic evaluations on it. If the complementary Neurostatus-form "SMARTCARE (smartly modernized assessment - recorded, telemedical, care professional-assisted, remotely evaluated)" was equal to the standard Neurostatus-EDSS, it could be applied at patients' homes in decentralized clinical trials or telemedical clinical consultations.

In this study the Neurostatus-SMARTCARE, performed by trained HCPs is compared to the standard Neurostatus-EDSS, performed by neurologists.

At two routine clinical visits a neurologist and a nurse perform the EDSS one after the other with a break for the patient as needed. To account for potential sequence effects, the order of assessment is randomly assigned to "first neurologist, then nurse" (group A) and "first nurse, then neurologist" (group B). At the next clinical consultation (visit 2), the reverse order is applied. All assessments are video-recorded.

Each pair of assessment is compared with regard to concordance as to the 3 levels of the scale: EDSS step, Functional System Scores (FSS) and subscores. Comparison is automated in a digital tool. In case of discrepancies, an EDSS expert assesses the videos to determine, which is the correct examination result.

The neurologists and nurses are blinded to each others' assessment results and to the participants' previous EDSS step. The experts are blinded to the raters' identity until the moment of watching a video.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old at the time of signing the informed consent
* Clinically definite MS, confirmed through the medical chart
* At least one documented EDSS assessment within two (2) years prior to inclusion
* The participant must be capable of giving signed informed consent

Exclusion Criteria:

* Insufficient knowledge of the German language, i.e. inability to understand the patient information or to follow the instructions and questions during the EDSS assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Inter-rater reliability, i.e. the concordance rate between Neurostatus-SMARTCARE and Neurostatus-EDSS® at EDSS step level | 1.5 - 2 hours per study visit for each participant
  The pairwise concordance among all EDSS-steps between a neurologist's and a nurse's assessment of the the same participant at one visit will be tested and an overall concordance rate of all EDSS-steps.
  The true concordance level needs to be at least 89% to have a reasonable chance of demonstrating that the observed rate is significantly higher than 80%. If this can be shown, it can be concluded that Neurostatus-SMARTCARE is equivalent to the standardized Neurostatus-EDSS in clinical routine or clinical trials. This would allow HCPs to assess the Neurostatus-EDSS with the same quality as neurologists.

SECONDARY OUTCOMES:
Inter-rater reliability at subscore level between Neurostatus-SMARTCARE and standard Neurostatus-EDSS® | 1.5 - 2 hours per study visit for each participant
  The pairwise concordance among all subscores between a neurologist's and a nurse's assessment of the the same participant at one visit will be tested and an overall concordance rate of all subscores.
Inter-rater reliability at Functional System Score (FSS) levels between Neurostatus-SMARTCARE and standard Neurostatus-EDSS® | 1.5 - 2 hours per study visit for each participant
  The pairwise concordance among all FSS between a neurologist's and a nurse's assessment of the the same participant at one visit will be tested and an overall concordance rate of all FSS.
Number of assessments rated correctly by neurologists in comparison to HCPs | Through study completion, an average of 1.5 years
  When discrepancies occur between neurologists and nurses at EDSS step level, it will be calculated how often the neurologists had assessed the correct result and how often the nurses.
Number and type of the same error occurring more than once at the individual rater level | Through study completion, an average of 1.5 years
  It will be tested if raters make the same error more than once, i.e. if they make typical errors that could be corrected through re-training. Therefore the number of "more-than-once-errors" will be collected and the type of error, e.g. errors through a false examination technique or a calculation error in determining the FSS/ EDSS step.
Inter-rater reliability in capturing the number of changes in the Expanded Disability Status Scale (EDSS) through worsening and progression or improvement occurring between the first and second measurement. | Through study completion, an average of 1.5 years
  I twill be tested if neurologists and nurses detect EDSS changes after 6 months equally, i.e. if they assign the same changed EDSS step.
  Note: Changes in the EDSS are defined in steps of 0.5 points. Increasing numbers of the EDSS step mean worsening, decreasing numbers mean improvement. An increase of 1.0 point over 3 months is usually considered MS progression.

CONTACTS AND LOCATIONS:
Overall Officials: Ludwig Kappos, Prof. Dr. med. Dr. h. c. mult., Study Director — Foundation Clinical Neuroimmunology and Neuroscience Basel (RC2NB)
Locations (2):
- Switzerland (2):
  - Neurologic Clinic and Policlinic, University Hospital Basel, Basel
  - Luzerner Kantonsspital, Lucerne